CLINICAL TRIAL: NCT04074967
Title: A Phase Ib/II Study of ARRY-614 Plus Either Nivolumab or Nivolumab+Ipilimumab in Advanced Solid Tumors
Brief Title: Study of ARRY-614 Plus Either Nivolumab or Nivolumab+Ipilimumab
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 19-097
Record Dates: First submitted 2019-08-19; First posted 2019-08-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Melanoma; Solid Tumor; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase lb: subjects with advanced solid tumors will receive ARRY-614 in combination with nivolumab or ARRY-614 in combination with nivolumab + ipilimumab immunotherapy.
  Phase ll: Subjects with NSCLC or HNSCC will receive ARRY-614 combined with nivolumab. Subjects with melanoma will receive ARRY-614 combined with nivolumab + ipilimumab. Subjects with RCC will receive ARRY-614 combined with nivolumab + ipilimumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase Ib ARRY-614 + nivolumab (Experimental): Participants with advanced solid tumors will receive ARRY-614 in combination with nivolumab.
  (histologically confirmed metastatic or unresectable malignancy with lacking curative measures; nivolumab must be available and appropriate for proposed therapy)
  Interventions: Drug: Phase Ib ARRY-614 + nivolumab
- Phase Ib ARRY-614 + nivolumab + ipilimumab (Experimental): Participants with advanced solid tumors will received ARRY-614 in combination with nivolumab + ipilimumab.
  (histologically confirmed metastatic or unresectable malignancy with lacking curative measures; nivolumab and ipilimumab must be available and appropriate for proposed therapy)
  Interventions: Drug: Phase Ib ARRY-614 + nivolumab+ipilimumab
- Phase II ARRY-614 + nivolumab (Experimental): Participants with of NSCLC and HNSCCC will receive ARRY-614 combined with nivolumab.
  Interventions: Drug: Phase II ARRY-614 + nivolumab
- Phase II ARRY-614 + nivolumab + ipilimumab (melanoma) (Experimental): Participants with melanoma will receive ARRY-614 combined with nivolumab + ipilimumab.
  Interventions: Drug: Phase II ARRY-614 + nivolumab+ipilimumab (melanoma)
- Phase II ARRY-614 + nivolumab + ipilimumab (RCC) (Experimental): Participants with RCC will receive ARRY-614 combined with nivolumab + ipilimumab.
  Interventions: Drug: Phase II ARRY-614 + nivolumab+ipilimumab (RCC)

INTERVENTIONS:
Drug: Phase Ib ARRY-614 + nivolumab — ARRY-614 continuously in 4-week cycles (± 3 days). Nivolumab will be dosed according to FDA-approved dosing schedule.
  Arms: Phase Ib ARRY-614 + nivolumab
Drug: Phase Ib ARRY-614 + nivolumab+ipilimumab — ARRY-614 continuously in 4-week cycles (± 3 days). Nivolumab will be dosed according to FDA-approved dosing schedule. Ipilimumab therapy will be dosed according to FDA-approved dosing schedule.
  Arms: Phase Ib ARRY-614 + nivolumab + ipilimumab
Drug: Phase II ARRY-614 + nivolumab — Recommended Phase II dose of ARRY-614 (to be determined) daily in 4-week cycles (± 3 days).
  Nivolumab will be dosed according to FDA-approved dosing schedule.
  Arms: Phase II ARRY-614 + nivolumab
Drug: Phase II ARRY-614 + nivolumab+ipilimumab (melanoma) — Recommended Phase II dose of ARRY-614 (to be determined) daily in 4-week cycles (± 3 days).
  Nivolumab will be dosed according to FDA-approved dosing schedule. Ipilimumab therapy will be dosed according to FDA-approved dosing schedule.
  Arms: Phase II ARRY-614 + nivolumab + ipilimumab (melanoma)
Drug: Phase II ARRY-614 + nivolumab+ipilimumab (RCC) — Recommended Phase II dose of ARRY-614 (to be determined) daily in 4-week cycles (± 3 days).
  Nivolumab will be dosed according to FDA-approved dosing schedule. Ipilimumab therapy will be dosed according to FDA-approved dosing schedule.
  Arms: Phase II ARRY-614 + nivolumab + ipilimumab (RCC)

SUMMARY:
In this study, the Phase Ib portion aims to establish safety and tolerability of ARRY-614 with either nivolumab or ipilimumab and to determine a recommended phase II dose of ARRY-614 in combination with either nivolumab or nivolumab+ipilimumab immunotherapy in patients with selected advanced solid tumors. The Phase II portion will estimate the efficacy of ARRY-614 in combination with either nivolumab or ARRY-614 + nivolumab+ipilimumab immunotherapy in patients with with NSCLC, HNSCC, melanoma and RCC and melanoma.

DETAILED DESCRIPTION:
This phase Ib/II study of PO administered ARRY-614 in combination with checkpoint immunotherapy. In phase Ib, this includes ARRY-614 plus nivolumab or ARRY-614 + nivolumab+ipilimumab in patients with selected advanced solid tumors. In phase II, this includes ARRY-614 in combination with nivolumab in a combined cohort of NSCLC and HNSCCC as well as two arms with patients having either melanoma and RCC, where ARRY-614 will be combined with nivolumab+ipilimumab. The objective of the Ib phase is to determine the safety, tolerability and recommended phase II dose of ARRY-614 with either nivolumab or nivolumab+ipilimumab combination therapy. The objective of Phase II is to determine best ORR in the three separate phase II arms: ARRY-614 plus nivolumab+ipilimumab in melanoma or RCC as well as ARRY-614 plus nivolumab in a combined cohort of NSCLC and HNSCC. The recommended phase II dose will be informed by the phase Ib safety study of ARRY-614, the plasma PK of ARRY-614 and the metabolite, AR00451575, and the PD effects of ARRY-614 in pre and post dose peripheral blood samples.

In phase Ib, trial participants will take ARRY-614 continuously in 3- or 4-week cycles (± 3 days). Nivolumab and nivolumab+ipilimumab therapy will be dosed according to FDA-approved or compendium supported dosing schedule.

In phase II, a similar dosing schedule will be pursued once the recommended phase II dose of ARRY-614 has been determined with nivolumab or nivolumab +ipilimumab. ARRY-614 will be given on a daily PO schedule in 3- or 4-week cycles (± 3 days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* For Phase Ib: Trial participants must have a histologically confirmed malignancy that is metastatic or unresectable for which curative measures do not exist or are no longer effective.

  a.Trial participants must have nivolumab or ipilimumab therapy available and must be appropriate for this therapy.
* For Phase II:

  1. Participants with melanoma who previously experienced disease progression on anti-PD1 (with or without ipilimumab).
  2. Participants with RCC who previously experienced disease progression on anti-PD1 (with or without ipilimumab).
  3. Participants with NSCLC or HNSCC who previously experienced disease progression on anti-PD1 (with or without ipilimumab).
  4. Progression on prior anti-PD1/L1 or anti-PD1/anti-CTLA4 antibodies must meet definitions for primary or secondary resistance and regrowth after stopping therapy as below or there must be documentation by the treating investigator of rapid disease progression such that these criteria cannot be assessed (suggestions from the Society for ImmunoTherapy of Cancer PD1 Resistance Working Group).
* Have an ECOG PS score of 0 or 1 (Appendix 13.A).
* Have an expected survival of ≥3 months.
* Have at least one evaluable and measurable lesion as defined by RECIST v1.1.
* The first five patients in each Phase II cohort must have tumors determined to be easily accessible for biopsy and must be willing to have two biopsies
* Have recovered from toxicities associated with prior anticancer therapy to baseline or Grade 1 unless stabilized under medical management per investigator.
* Have adequate bone marrow function as evidenced by:

  1. Absolute neutrophil count ≥1,500/mm3 or 1.5 ×109/L
  2. Hemoglobin ≥8 g/dL
  3. Platelets ≥100,000/mm3 or 100 × 109/L
* Have adequate hepatic function as evidenced by:

  1. Serum total bilirubin ≤2 × upper limit of normal (ULN), unless considered due to Gilbert's disease
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x the institutional ULN or ≤ 5.0x institutional ULN in the presence of known liver metastases.
* Patients with creatinine clearance > 30 mL/min, (measured using Cockcroft-Gault equation or the estimated glomerular filtration rate from the Modification of Diet in Renal Disease Study) are included in the study.
* Be able to understand and willing to sign the informed consent form (or have legal representation) and to comply with scheduled visits, treatment plans, procedures, and laboratory tests, including serial peripheral blood sampling, biopsies, and urine sampling, during the study. A legally authorized representative may consent on behalf of a subject who is otherwise unable to provide informed consent if acceptable to and approved by the site's IRB/Independent Ethics Committee (IEC).
* Female patients with reproductive potential must have a negative serum pregnancy test prior to the start of therapy, or a confirmation from an obstetrician in case of equivocal serum pregnancy results. Females of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion or who have not been naturally postmenopausal (ie, who have not menstruated) for at least 24 consecutive months (ie, have not had menses at any time in the preceding 24 consecutive months). Women with reproductive potential, as well as fertile men and their partners who are female with reproductive potential, must agree to use two effective forms of contraception (including at least one barrier form) from the time of giving informed consent throughout the study and for 5 months after the last dose of therapy for women, and 7 months after last dose for men. Effective forms of contraception are defined as hormonal PO contraceptives, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization.
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  1. A stable regimen of highly active anti-retroviral therapy (HAART)
  2. No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  3. A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based test

Exclusion Criteria:

* Received systemic anticancer therapy or an investigational agent <2 weeks prior to Day 1 (washout from prior immune based anticancer therapy is 4 weeks). In addition, the first dose of study treatment should not occur before a period ≥5 half-lives of the investigational agent has elapsed (excluding nivolumab therapy or combination anti-PD1/ipilimumab combination therapy in RCC - prior ipilimumab not permitted in melanoma cohort).
* For ST, have underwent hepatic radiation, chemoembolization, and radiofrequency ablation <4 weeks prior to Day 1.
* Participants must not have had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 (with exception of anti-PD1/ipilimumab combination therapy) or have not recovered (i.e. < Grade 1 at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Participants must not have a diagnosis of immunodeficiency or be receiving systemic steroid therapy at a dose of >10 mg prednisone daily or equivalent at time of first dose of trial treatment (this criterion does not apply to HIV-positive patients as detailed in the inclusion criteria).
* Participants must not have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Participants must not have a known history of non-infectious pneumonitis that required steroids for treatment.
* Participants must not have evidence of active interstitial lung disease.
* Have known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 1 week and have radiographically stable disease for at least 1 month prior to study entry. Note: up to 10 mg per day of prednisone equivalent will be allowed.
* Have a history of another primary cancer that is active requiring treatment, progressing or for which the investigator believes will make disease assessment unreliable.
* Underwent major surgery within 4 weeks of Day 1 or have not recovered from post-surgery toxicities.
* Are pregnant or breastfeeding.
* Have an active infection requiring systemic anti-infective therapy or with an unexplained fever >38.5°C within 7 days of Day 1 (at the discretion of the Investigator, patients with tumor fever may be enrolled).
* Have any known hypersensitivity to any of the components of ARRY-614 or anti-PD1/ipilimumab combination therapies.
* Have significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) Class III or IV congestive heart failure); myocardial infarction; unstable angina; and/or stroke.
* Have known LVEF <40% by ECHO scan (or by other methods according to institutional practice) obtained within 28 days prior to the start of study treatment (testing is not otherwise mandatory).
* Have known active hepatitis B (HBV) or hepatitis C (HCV) infections. Patients with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Patients with chronic HBV that is adequately suppressed per institutional practice will be permitted.
* Have any other acute or chronic medical or psychiatric condition, including recent (within 12 months of Day 1) or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
* Have known active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered PO. Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential).
* Have been committed to an institution by an order issued either by the judicial or administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants Experiencing a Dose Limiting Toxicity (DLT) | Up to 28 days (during first cycle of treatment)
  Safety and recommended Phase ll dose of ARRY-614 in combination with either nivolumab or or nivolumab+ipilimumab per NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.0: Any AE (unless attributable to an extraneous cause, ex. disease progression) that satisfies ≥1 of the following: Grade 3 or 4 nausea or vomiting; Grade 3 or 4 nausea or vomiting despite anti emetic prophylaxis; Grade 3 or 4 diarrhea; Grade 3 or 4 diarrhea despite the administration of anti-diarrheals. Other Grade 3 or 4 (except asymptomatic amylase/lipase or other asymptomatic biochemical marker that does not resolve with adequate treatment in ≤1 week). Hematologic AEs: Absolute neutrophil count (ANC) <500/mm^3 for ≥5 days, Febrile neutropenia (ANC < 1,000/mm^3 and single temperature ≥38.3 °C or sustained temperature of ≥38.0 °C for ≥1 hour), Platelets <25,000/mm^3, Hemoglobin <8.0 g/dL, Grade 3 hemorrhage associated with thrombocytopenia < Grade 4 (i.e. Grade 3 hemorrhage with platelets >25,000/mm^3).
Objective Response | Up to 48 months
  The probability of (objective) response to treatment (estimation). Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

SECONDARY OUTCOMES:
Adverse Events related to Study Treatment | Up to 48 months
  The occurrence (number and type) of toxicity events in participants receiving ARRY-614 in combination with either nivolumab or or nivolumab+ipilimumab immunotherapy. Adverse Events and Serious Adverse Events per CTCAE v5.0 at least Possibly Related to Treatment at (Phase II dose).
Overall Survival (OS) | Up to 48 months
  The length of time from the start of treatment that diagnosed participants remain alive, until the time of death from any cause.
Progression Free Survival (PRS) | Up to 48 months
  The length of time from first dose of either drug until disease progression or death from any cause, whichever occurs first.Per RECIST v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Duration of Response | Up to 48 months
  Time between the initial response to treatment per RECIST v1.1 and subsequent disease progression.
  Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Response per Immune-related response criteria (irRECIST) | Up to 48 months
  irCR (Complete Response):Disappearance of non-nodal lesions.All pathologic lymph nodes <10 mm (2 consecutive measures ≥4 weeks apart); irPR (Partial Response):≥30% decrease from baseline (2 consecutive measures ≥4 weeks apart); irPD (Progressive Disease):≥20% increase from nadir and ≥5mm (2 consecutive measures ≥4 weeks apart); irSD (Stable Disease): Not sufficient decrease for PR, nor sufficient increase for PD; irPR (Progressive Disease): Disappearance of all non-nodal lesions.All pathologic lymph nodes <10 mm (Non-Target Lesions:Any other than disappearance of all non-nodal lesions and reduction of pathologic lymph nodes <10 mm). Baseline tumor burden: sum of single diameters (short axis for nodal lesions, longest diameter for other lesions) for target lesions. In subsequent scans, the diameters of new measurable lesions are added to the tumor burden. Re-treatment: ≤5 target lesions (=/≠ original lesions) are selected and a new baseline tumor burden will be established.

OTHER OUTCOMES:
Pharmacokinetic profile of ARRY-614 | Day 1 and 15 of Cycle 1, Day 1 and 15 of Cycle 2, and Day 1 of subsequent cycles (28 day cycles); up to 3 months
  Plasma concentrations and PK for ARRY-614 and its metabolite potentially, including Maximum Plasma Concentration [Cmax].
Tumor Inflammation Signature (TIS) score | 28 days prior to treatment, Day 1 of Cycle 1, Cycle 2 and subsequent cycles (28 day cycles); up to 3 months
  The Tumor Inflammation Signature (TIS) is an investigational use only (IUO) 18-gene signature that measures a pre-existing but suppressed adaptive immune response within tumors using a gene expression algorithm. Higher TIS scores are associated with an increase in overall response rate and better prognosis.
Pharmacodynamic profile of ARRY-614 | 28 days prior to treatment, Days 1 and 15 of Cycles 1 and 2, and Day 1 of Cycle 3; up to 3 months
  Gene expression changes will be presented as either positive (+) or negative (-).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No